CLINICAL TRIAL: NCT04252105
Title: The Effect of an Antioxidant-rich Kindergarten Diet on Oxidative Stress in Healthy Preschool Children
Brief Title: Antioxidant-rich Diet and Oxidative Stress in Healthy Preschoolers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana, Faculty of Medicine (Other)
Collaborators: University of Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Ox-Stress-Preschool
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Oxidative Stress
MeSH Terms: interventions — Antioxidants

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antioxidant rich diet (Experimental)
  Interventions: Dietary Supplement: Antioxidant
- Regular diet (No Intervention)

INTERVENTIONS:
Dietary Supplement: Antioxidant — Antioxidant-rich diet (added selected types of fruits, vegetables, nuts, cereals and oils)
  Arms: Antioxidant rich diet

SUMMARY:
Uncontrolled and prolonged oxidative stress plays an important role in the onset and progression of cardiovascular disease, hyperlipidemia, diabetes, and various cancers. Given that many diseases can start as early as childhood, eating patterns in childhood and preventing oxidative damage can have beneficial long-term health effects. Antioxidant-rich foods can slow down the progression of chronic diseases.

In Slovenian kindergartens (and schools) children consume up to 70% of their daily energy and nutritional needs, so what is offered to them is very important. This study will evaluate the hypothesis that providing an antioxidant-rich diet in kindergartens can result in the reduction of biomarkers of oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* • Healthy children aged 5-6 who will attend the compulsory medical examination before entering primary school

Exclusion Criteria:

* • Children with chronic conditions (e.g. diabetes, asthma)

  * Children with allergies to food (e.g. gluten, egg, milk, lactose intolerance)

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Oxidative stress biomarkers | 2 weeks
  Change in oxidative stress biomarkers of lipids (malondialdehyde (MDA), and four F2 - isoprostane isomers, namely 8 -iso-prostaglandin F2α (8-PGF2α), 11ß- prostaglandin F2α (11-PGF2α), 15 (R)-prostaglandin F2α (15-PGF 2α) and 8-iso, 15 prostaglandin F2α (8,15-PGF2α) ; proteins (o,o'-dityrosine (diY) and DNA 8-Hydroxy-2'-deoxyguanosine (8-OhdG) between day 1 and day 15 of the intervention diet, measured by HPLC-MS/MS

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ljubljana, Faculty of Medicine, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Berlic M, Korosec M, Remec ZI, Cuk V, Battelino T, Repic Lampret B. Effect of antioxidant-rich kindergarten meals on oxidative stress biomarkers in healthy 5-6-year-old children: a randomized controlled trial. Eur J Pediatr. 2024 Jul;183(7):3085-3094. doi: 10.1007/s00431-024-05576-6. Epub 2024 Apr 25. PMID 38658398